CLINICAL TRIAL: NCT04654949
Title: Pilot Pragmatic Randomized Controlled Trial: The Effects of Horticultural Therapy (HT) vs Existing Care on Engagement, Mood and Mobility of Inpatient Older Adults in an Acute Care Hospital
Brief Title: Pilot Pragmatic Randomized Controlled Trial: Horticultural Therapy for Inpatient Older Adults in an Acute Care Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/00211
Record Dates: First submitted 2020-10-27; First posted 2020-12-04 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Frailty; Hospitalism
Keywords: Horticultural Therapy; Randomized controlled trial
MeSH Terms: conditions — Frailty | interventions — Horticultural Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horticultural Therapy (Experimental): The Horticultural Therapy group receives 30 minutes of horticultural therapy activities using mobile horticulture kits conducted by therapists or therapy assistants to engage participants at their bedside.
  Interventions: Other: Horticultural Therapy
- Existing Care (No Intervention): The existing Care group receives 30 minutes of routine ward-based engagement leisure activities (e.g. watching television, reading newspapers, etc).

INTERVENTIONS:
Other: Horticultural Therapy — The horticultural therapy sessions are conducted by the occupational therapists or therapy assistants using the mobile horticultural kits. The horticultural activities are designed to stimulate the senses through interaction with specific tasks and the environment, promote social interaction, mobility and also promote a sense of self-worth through various horticultural activities such as planting seeds, transplanting plants, trimming and watering plants.
  Arms: Horticultural Therapy

SUMMARY:
This study aims to investigate the feasibility and effectiveness of Horticultural Therapy (HT) on engagement, mood, and quality of life (QoL) of older adults in geriatric acute care in Singapore. Investigators will also assess the effectiveness of HT on mobility and hospitalisation experience. This pilot study could inform how HT can be implemented in geriatric acute care and its effect on hospitalisation experience and recovery of function.

DETAILED DESCRIPTION:
Horticultural therapy (HT) is a non-pharmacological treatment utilizing plant-related activities as a form of alternative medicine to achieve specific goals that lead to person's well-being. Geriatric patients in acute care wards are at risk of functional decline related to acute illness and prolonged bed rest during hospitalization. HT can complement medical treatment to ameliorate the adverse effects of hospitalisation in older adults. There is evidence that HT can improve the physical and psychological well-being of the older adults in different settings. The beneficial effects of HT have mostly been documented in nursing homes, community rehabilitation facilities and senior activity centres, but not in geriatric acute care settings. There is also a need to harness available knowledge and implement it where appropriate. This study aims to investigate the feasibility and effectiveness of HT on engagement, mood, and quality of life (QoL) of older adults in geriatric acute care in Singapore. Investigators will also assess the effectiveness of HT on mobility and hospitalisation experience. This pilot study could inform how HT can be implemented in geriatric acute care and its effect on hospitalisation experience and recovery of function.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old and above
* an inpatient in Khoo Teck Puat Hospital
* able to understand simple instructions (with abbreviated mental test's score of 6 and above)
* have stable vital signs - blood pressure, heart rate and peripheral capillary oxygen saturation - to take part in horticultural therapy activities

Exclusion Criteria:

* on contact or droplet precaution
* diagnosed with severe auditory-visual impairments
* have major depressive disorder
* have endocrine disorders
* on steroid-based medications such as asthma and allergies that might affect the salivary cortisol level
* on the Dangerously Ill List

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Average Score of Engagement Assessed by Menorah Park Engagement Scale (MPES) | Five days
  MPES consists of four different types of engagement: "constructive", "passive", "self" and "none" (Judge, Camp & Orsulic-Jeras, 2000).
  Each type of engagement is recorded on five-minutes intervals during the 30-minutes sessions for both intervention and control group. The score of 0, 1 and 2 represent engagement "not observed", "observed for less than two and a half minutes" and "observed for more than two and a half minutes" respectively.
  The average score of each type of engagement for all sessions during assessment period is compared between the two groups. The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.
Average Score of Mood Assessed by Apparent Affect Rating Scale (AARS) | Five days
  AARS consists of five different domains of mood: pleasure, general alertness, anxiety/ fear, anger and sadness (Lawton, Haitsma & Klapper, 1996).
  Each domain of mood is recorded on five-minutes intervals during the 30-minutes sessions for both intervention and control group. The score of 0, 1 and 2 represent engagement "not observed", "observed for less than two and a half minutes" and "observed for more than two and a half minutes" respectively.
  The average score of each domain of mood for all sessions during assessment period is compared between the two groups. The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.
Change in Mobility Performance Assessed by Modified Perme ICU scale | Five days
  Change in mobility performance from baseline (before randomization) to last session during the assessment period is measured by the modified Perme ICU scale (Perme, Nawa, Winkelman & Masud, 2014).
  The mobility domains of "bed mobility", "transfers" and "gait" are recorded with the score of 0 to 7, indicates for "total assistance", "maximum assistance", "moderate assistance", "minimal assistance", "contact guard", "standby assistance", "supervision" and "independent" respectively.
  The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.
Change in Quality of Life Assessed by the EQ-5D | Five days
  Change in quality of life is measured by the change in the score of the EuroQol EQ-5D from baseline (before randomization) to last session during the assessment period (Brooks & Charro, 1996). The EQ-5D covers five dimensions on health status - mobility, self-care, usual activities and anxiety/depression using 5 response levels - no problem, slight problem, moderate problem, severe problem and extreme problem.
  The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.

SECONDARY OUTCOMES:
Number of Transitions in the Mobility Status | Five days
  Participants' mobility state at the start of the session, the highest mobility state during session and the number of transitions in the mobility are captured using the mobilisation scale. The average score of highest mobility status and number of transitions in the mobility are compared between intervention and control group. The higher the score indicates better outcome.
  The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.
Change in Emotion Assessed by Emoticon Scale | 5 days
  The Emoticon Scale consists of seven simple emotion icons with smiling faces (A/1-C/3), a neutral face (D/4), and frowning faces (E/5-G/7) on a Likert scale (Tan et al., 2018). Participants are asked to rate their mood at point of assessment at baseline (before randomisation) and at the last session of the assessment period.
  The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.
Hospitalisation Experience Questionnaire | Five days
  It is a 10-self administered questionnaire modified from the Person-centered care assessment tool (PCAT) (Edvardsson et al., 2010) which aims to evaluate the quality of health care settings as perceived by patients.
  The score is Likert scale from 0 to 5, with 0 indicating "No, I disagree completely" and 5 indicating "Yes, I agree completely". Hospitalisation Experience Questionnaire is administered at the last session of the assessment period.
  The assessment period is five days, or from recruitment date to participants' discharge date from the acute care hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Thuy-Anh Giang, Principal Investigator — Khoo Teck Puat Hospital
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

REFERENCES:
- [Background] Nicholas SO, Giang AT, Yap PLK. The Effectiveness of Horticultural Therapy on Older Adults: A Systematic Review. J Am Med Dir Assoc. 2019 Oct;20(10):1351.e1-1351.e11. doi: 10.1016/j.jamda.2019.06.021. Epub 2019 Aug 8. PMID 31402135